CLINICAL TRIAL: NCT04375046
Title: Recombinant Bacterial ACE2 Receptors -Like Enzyme of B38-CAP Could be Promising Treatment for COVID-19 Infection- and Its Inflammatory Complications Better Than Recombinant Human ACE2
Acronym: Bacterial ACE2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: proposed by Mahmoud kazazzaz
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID 2019 ,Infection, B38-CAP , Bacterial ACE2 receptors -like enzyme , rhACE226
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: rbACE2 group (Experimental): 0.4 mg/kg IV BID for 7 days (unblinded) + standard of care
  Interventions: Drug: Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP (rbACE2)
- No Intervention: Control group (No Intervention): Standard of care; no placebo

INTERVENTIONS:
Drug: Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP (rbACE2) — In this study, the experimental group will receive 0.4 mg/kg rbACE2 IV
  Arms: Experimental: rbACE2 group

SUMMARY:
Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP could be promising treatment for COVID-19 infection- and Its inflammatory complications better than recombinant human ACE2

Mahmoud ELkazzaz(1),Tamer Haydara(2),Yousry Abo-amer(3), Quan Liu(4)

1. Department of chemistry and biochemistry, Faculty of Science, Damietta University, Egypt.
2. Department of Internal Medicine, Faculty of Medicine, Kafrelsheikh University, Egypt
3. Hepatology,Gastroenterology and Infectious Diseases Department, Mahala Hepatology Teaching Hospital, Egypt
4. School of Life Sciences and Engineering, Foshan University, Foshan, Guangdong Province; Laboratory of Emerging Infectious Disease, Institute of Translational Medicine, The First Hospital of Jilin University, Changchun, China.

Abstract

The COVID-19 pandemic caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has infected over 100 million people causing over 2.4 million deaths over the world, and it is still expanding. There is an urgent need for targeted and effective COVID-19 treatments which has put great pressure on researchers across the world for developing effective drugs. This paper reviews the possibility of using Recombinant Bacterial ACE2 Receptors -Like Enzyme of B38-CAP to treat SARS-CoV-2 based on the intracellular mechanism of SARS-CoV-2 transmission and consequences caused. Angiotensin-converting enzyme 2 (ACE2) plays a key role in cardiovascular physiology and pathology, and it's being currently being investigated as a potential covid-19 and acute lung failure treatment through several clinical trials.. The SARS-CoV2 binding site was identified as ACE2, a part of the RAAS, which is known to protect the lung from injuries. it has been postulated that SARS-CoV-2 binding to ACE2 may attenuate residual ACE2 activity, skewing the ACE/ACE2 balance to a state of heightened angiotensin II activity leading to inflammatory and oxidative organ damage, as well as pulmonary vasoconstriction, which can lead to acute lung injury.. Therefore, treatment with recombinant soluble ACE2 protein and drugs that up regulate ACE2 may alleviate pulmonary complication. In animal models including heart failure, acute lung injury, and diabetic nephropathy, recombinant human ACE2 protein (rhACE2), which is devoid of its membrane-anchored domain thus soluble, has been shown to have beneficial effects. Despite its positive effects, rhACE2 is a glycosylated protein, which necessitates a time- and cost-intensive protein expression system using mammalian or insect cells, which may be inconvenient in drug production and medical economics. Moreover, we hypothesis that treating COVID-19 patients with recombinant soluble ACE2 protein may induce autoantibodies and T cells to cellular ACE2.Furthermore, rhACE2 may interact with spike protein based vaccine and worsen its effect . These autoantibodies may generated by enforced presentation of the soluble Angiotensin-converting enzyme 2 (ACE2) protein in a complex with COVID-19 Spike protein in fragment crystallizable (FC) Receptor positive Antigen Presenting Cells in the blood The development of autoantibodies might make injury and damage to the host epithelial cells and hamper their ACE2 dependent function in lungs, intestine and testes which express ACE2. In addition to inducing platelet aggregation and thrombosis . Although it has been stated that immune response associated with the chronic infusion of rhACE2 resulting in the degradation of rhACE226, this was not the case with B38-CAP; no antibodies against B38-CAP were detected in the serum of mice infused with B38-CAP for two weeks... In this case we suggest that bacterial engineering could be used to develop better protein drugs for COVID-19 treatment... B38-CAP is an ACE2-like enzyme derived from bacteria that reduces hypertension and cardiac dysfunction. Angiotensin-converting enzyme 2 (ACE2) plays a key role in cardiovascular physiology and pathology, and it is currently being studied in clinical trials to treat acute lung failure. In mice, B38-CAP treatment prevented angiotensin II-induced hypertension, cardiac hypertrophy, and fibrosis. B38-CAP is an ACE2-like enzyme derived from bacteria, demonstrating that evolution has shaped a bacterial carboxypeptidase (B38-CAP) to a human ACE2-like enzyme. As a result, we think that treating COVID-19-infected patients with Bacterial ACE2 like enzymes, rather than human ACE2, may be preferable because it will perform the same role as human ACE2 and may not be recognized by COVID-19 spike protein

Keywords: COVID 2019 ,Infection, B38-CAP , Bacterial ACE2 receptors -like enzyme , rhACE226.

DETAILED DESCRIPTION:
Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP could be promising treatment for COVID-19 infection- and Its inflammatory complications better than recombinant human ACE2

This is a small pilot study investigating whether there is any efficacy signal that warrants a larger Phase 2B trial, or any harm that suggests that such a trial should not be done. It is not expected to produce statistically significant results in the major endpoints. The investigator will examine all of the biologic, physiological, and clinical data to determine whether a Phase 2B trial is warranted.

Primary efficacy analysis will be carried only on patients receiving at least 4 doses of active drug. Safety analysis will be carried out on all patients receiving at least one dose of active drug.

It is planned to enroll more than or equal to 24 subjects with COVID-19. It is expected to have at least 12 evaluable patients in each group.

Experimental group: 0.4 mg/kg rbACE2 IV BID and standard of care Control group: standard of care Intervention duration: up to 7 days of therapy No planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory diagnosis:

   Respiratory specimen is positive for SARS-CoV-2 nucleic acid by RT-PCR; OR, The viral gene sequencing of the respiratory specimen is highly homologous to known novel coronavirus.
2. Fever:

   Axillary temperature >37.3℃
3. Respiratory variables (meets one of the following criteria):

   * Respiratory rate: RR ≥25 breaths/min
   * Oxygen saturation ≤93% at rest on room air
   * PaO2/FiO2 ≤300 mmHg（1 mmHg=0.133 KPa）
   * Pulmonary imaging showed that the lesions progressed more than 50% within 24-48 hours, and the patients were managed as severe
4. HBsAg negative, or HBV DNA ≤10^4 copy/ml if HBsAg positive; anti-HCV negative; HIV negative two weeks prior to signed Informed Consent Form (ICF)
5. Appropriate ethics approval and
6. ICF -

Exclusion Criteria:

* Age <18 years; Age >80 years
* Pregnant or breast feeding woman or with positive pregnancy test result P/F <100 mmHg
* Moribund condition (death likely in days) or not expected to survive for >7 days Refusal by attending MD
* Not hemodynamically stable in the preceding 4 hours (MAP ≤65 mmHg, or SAP <90 mmHg, DAP <60 mmHg, vasoactive agents are required)
* Patient on invasive mechanical ventilation or ECMO
* Patient in other therapeutic clinical trial within 30 days before ICF
* Receive any other ACE inhibitors (ACEI), angiotensin-receptor blockers (ARB) treatment within 7 days before ICF
* Chronic immunosuppression: current autoimmune diseases or patients who received immunotherapy within 30 days before ICF
* Hematologic malignancy (lymphoma, leukemia, multiple myeloma)
* Other patient characteristics (not thought to be related to underlying COVID-19) that portend a very poor prognosis (e.g, severe liver failure, and ect)
* Known allergy to study drug or its ingredients related to renin-angiotensin system (RAS), or frequent and/or severe allergic reactions with multiple medications
* Other uncontrolled diseases, as judged by investigators
* Body weight ≥85 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Time course of body temperature (fever) | 14 days
  Compare the time course of body temperature (fever) between two groups over time.
Viral load over time | 14 days
  Compare viral load between two groups over time.

SECONDARY OUTCOMES:
P/F ratio over time | 14 days
  PaO2/FiO2 ratio
Sequential organ failure assessment score(SOFA score) over time | 14 days
  SOFA, including assessment of respiratory, blood, liver, circulatory, nerve, kidney, from 0 to 4 scores in each systems, the higher scores mean a worse outcome.
Pulmonary Severity Index (PSI) | 14 days
Image examination of chest over time | 14 days
  Based on radiologist's assessment of inflammatory exudative disease, category as follows: significant improvement, partial improvement, no improvement, increase of partial exudation, significant increase in exudation, unable to judge.
Proportion of subjects who progressed to critical illness or death | 14 days
Time from first dose to conversion to normal or mild pneumonia | 14 days
T-lymphocyte counts over time | 14 days
C-reactive protein levels over time | 14 days
Angiotensin II (Ang II) changes over time | 14 days
Angiotensin 1-7 (Ang 1-7) changes over time | 14 days
Angiotensin 1-5 (Ang 1-5) changes over time | 14 days
Renin changes over time | 14 days
Aldosterone changes over time | 14 days
Angiotensin-converting enzyme (ACE) changes over time | 14 days
Angiotensin-converting enzyme 2 (ACE2) changes over time | 14 days
Interleukin 6 (IL-6) changes over time | 14 days
Interleukin 8 (IL-8) changes over time | 14 days
Soluble tumor necrosis factor receptor type II (sTNFrII) changes over time | 14 days
Plasminogen activator inhibitor type-1 (PAI-1) changes over time | 14 days
Von willebrand factor (vWF) changes over time | 14 days
Tumor necrosis factor-α (TNF-α) changes over time | 14 days
Soluble receptor for advanced glycation end products (sRAGE) changes over time | 14 days
Surfactant protein-D (SP-D) changes over time | 14 days
Angiopoietin-2 changes over time | 14 days
Frequency of adverse events and severe adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: M.Sc. Mahmoud Elkazzaz, M.Sc.Biochemistry, Principal Investigator — General Organization of Export and Import control system

IPD SHARING:
Plan to Share IPD: No